CLINICAL TRIAL: NCT04857710
Title: Chronic Effects of Wide-pulse Neuromuscular Electrostimulation on Neuromuscular and Functional Properties in Healthy Subjects
Acronym: ELECTRO-WP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20CH198; 2021-A00507-34 (Other: ANSM)
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers
Keywords: Wide-pulse; Training; Strength gain; Neuromuscular adaptations; Neuromuscular electrostimulation

STUDY DESIGN:
Intervention Model Description: Evaluating and comparing the force gains induced by 2 NMES training programs (CONV, WP) applied on knee extensors in healthy subjects for 6 weeks. Understanding the neuromuscular adaptations involved in these gains, as well as the functional benefit resulting from these improvements. To consolidate the benefit of NMES programs, a control (CONT) modality is used as a reference and is representative of a sedentary behaviour regularly observed in our populations. The CONV modality allows us to compare with the current clinical application and the majority of the literature on the adaptations induced by NMES training. Finally, the WP modality aims to assess the possible benefits linked to the use of wide-pulses during the application of NMES.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (CONT) (Active Comparator): A control (CONT) modality is used as a reference and is representative of a sedentary behaviour regularly observed in our populations
  Interventions: Device: Control (CONT) modality
- Conventional neuromuscular electrostimulation (CONV) (Experimental): The CONV (conventional) modality allows us to compare with the current clinical application and the majority of the literature on the adaptations induced by NMES (neuromuscular electrostimulation) training.
  Interventions: Device: Conventional neuromuscular electrostimulation (CONV NMES)
- Wide-pulse neuromuscular electrostimulation (WP) (Experimental): The use of wide-pulse (WP) stimulations allows, in addition to the direct activation of the muscle fibers, the use of sensory pathways. This more global solicitation of the neuromuscular system (i.e. information going back to the spinal cord and even to the brain) prejudges more nervous adaptations and therefore a greater functional benefit.
  Interventions: Device: Wide-pulse neuromuscular electrostimulation (WP NMES)

INTERVENTIONS:
Device: Wide-pulse neuromuscular electrostimulation (WP NMES) — The WP NMES program consists of electrical stimulation trains of 1000 symmetrical biphasic pulses (1 ms, 100 Hz). The duration of a train is of 10 s and the rest between trains is of 30 s. A WP NMES session includes 30 evoked contractions. The stimulation intensity is monitored online and adjusted to the highest tolerable by the subjects.During the stimulation, subjects are seated with the knee joint fixed a 60° angle. Three self-adhesive electrodes are placed over the right thigh. The positive electrodes, measuring 25 cm² (5 x 5 cm), are placed as close as possible to the motor point of the vastus lateralis and vastus medialis muscles. The negative electrode, measuring 50 cm² (10 x 5 cm), is placed 5-7 cm below the inguinal ligament. Electrical stimulations are delivered by a stimulator BioStim (Mazet Santé).
  Arms: Wide-pulse neuromuscular electrostimulation (WP)
Device: Conventional neuromuscular electrostimulation (CONV NMES) — The CONV NMES program consists of electrical stimulation trains of 500 symmetrical biphasic pulses (0.2 ms, 50 Hz). The duration of a train is of 10 s and the rest between trains is of 30 s (duty cycle: 1/3). A WP NMES session includes 30 evoked contractions. The stimulation intensity is monitored online and adjusted to the highest tolerable by the subjects.
  During the stimulation, subjects are seated with the knee joint fixed a 60° angle. Three self-adhesive electrodes are placed over the right thigh. The positive electrodes, measuring 25 cm² (5 x 5 cm), are placed as close as possible to the motor point of the vastus lateralis and vastus medialis muscles. The negative electrode, measuring 50 cm² (10 x 5 cm), is placed 5-7 cm below the inguinal ligament. Electrical stimulations are delivered by a stimulator BioStim (Mazet Santé).
  Arms: Conventional neuromuscular electrostimulation (CONV)
Device: Control (CONT) modality — Control (CONT) modality is used as a reference and is representative of a sedentary behaviour regularly observed in our populations.
  Arms: Control (CONT)

SUMMARY:
Neuromuscular electrostimulation (NMES) is a technique used in the clinical and training fields to increase the strength of a muscle group.The recent use of wide-pulse (WP) stimulations allows, in addition to the direct activation of the muscle fibers, the use of sensory pathways. This more global solicitation of the neuromuscular system (i.e. information going back to the spinal cord and even to the brain) prejudges more nervous adaptations and therefore a greater functional benefit. The first aim of this study is to evaluate and compare the force gains induced by 2 NMES training programs (CONV, WP) applied on knee extensors in healthy subjects for 6 weeks.The second aim is to understand the neuromuscular adaptations involved in these gains, as well as the functional benefit resulting from these improvements.

DETAILED DESCRIPTION:
Neuromuscular electrostimulation (NMES) is a technique used in the clinical and training fields to increase the strength of a muscle group. The conventional (CONV) parameters of NMES induces a direct activation of the muscle fibers located close to the stimulation electrodes. This means that the neuromuscular system is not fully solicited, which limits its adaptation. The recent use of wide-pulse (WP) stimulations allows, in addition to the direct activation of the muscle fibers, the use of sensory pathways. This more global solicitation of the neuromuscular system (i.e. information going back to the spinal cord and even to the brain) prejudges more nervous adaptations and therefore a greater functional benefit.

The first aim of this study is to evaluate and compare the force gains induced by 2 NMES training programs (CONV, WP) applied on knee extensors in healthy subjects for 6 weeks. The second aim is to understand the neuromuscular adaptations involved in these gains, as well as the functional benefit resulting from these improvements. To consolidate the benefit of NMES programs, a control (CONT) modality is used as a reference and is representative of a sedentary behaviour regularly observed in our populations. The CONV modality allows us to compare with the current clinical application and the majority of the literature on the adaptations induced by NMES training. Finally, the WP modality aims to assess the possible benefits linked to the use of wide-pulses during the application of NMES. A clinical transfer will then be envisaged to confirm the interest and benefits of this type of program. We hypothesise that nervous adaptations will be increased by the use of WP NMES, leading to greater gains in strength and functional benefits than with CONV NMES.

ELIGIBILITY:
Inclusion Criteria:

* Affiliates or beneficiaries of a social security scheme
* Having freely given their written consent

Exclusion Criteria:

* Disease or surgery resulting in a locomotor disorder, within 6 months prior to the study
* Chronic neurological, motor or psychic diseases
* Taking neuro-active substances likely to alter cortico-spinal excitability (hypnotics, antiepileptics, psychotropic drugs, muscle relaxants) for the duration of the study
* Contraindication to neuromuscular electrostimulation
* Contraindication to magnetic stimulation
* Participation at the same time in another interventional experiment or having participated in such a study within 30 days prior to this study
* Sports (>10 hours per week or strength training of the lower limbs)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Maximal voluntary contraction (MVC) of the knee extensor muscle measurement | week 6
  Maximal isometric force (maximal voluntary contraction, MVC) of the knee extensor muscle

SECONDARY OUTCOMES:
Voluntary activation measurement (%) | week 6
  The level of voluntary activation will be determined by the force increment obtained following stimulation performed during a condition of the muscle in a state of maximum contraction.
Voluntary activation measurement (%) | week 12
  The level of voluntary activation will be determined by the force increment obtained following stimulation performed during a condition of the muscle in a state of maximum contraction.
Cortico-spinal excitability measurement | week 6
  The quantification of cortico-spinal excitability (i.e. motor evoked potentials, in mV) will be evaluated by recording the electromyographic responses (surface EMG) evoked by transcranial magnetic stimulation
Cortico-spinal excitability measurement | week 12
  The quantification of cortico-spinal excitability (i.e. motor evoked potentials, in mV) will be evaluated by recording the electromyographic responses (surface EMG) evoked by transcranial magnetic stimulation
Spinal excitability measurement | week 6
  The quantification of spinal excitability (i.e. spinal reflex, in mV) will be evaluated by recording the EMG responses evoked by electrical stimulation in the lumbar vertebrae.
  The quantification of spinal excitability (i.e. spinal reflex, in mV) will be evaluated by recording the EMG responses evoked by electrical stimulation in the lumbar vertebrae.
Spinal excitability measurement | week 12
  The quantification of spinal excitability (i.e. spinal reflex, in mV) will be evaluated by recording the EMG responses evoked by electrical stimulation in the lumbar vertebrae.
  The quantification of spinal excitability (i.e. spinal reflex, in mV) will be evaluated by recording the EMG responses evoked by electrical stimulation in the lumbar vertebrae.
Muscular endurance measurement | week 6
  Muscle endurance (number of contractions performed before failure) will be assessed during a fatigue protocol consisting of performing quadriceps muscle contractions at incremental strength levels.
Muscular endurance measurement | week 12
  Muscle endurance (number of contractions performed before failure) will be assessed during a fatigue protocol consisting of performing quadriceps muscle contractions at incremental strength levels.
Jump performances measurement | week 6
  The performance of jumps (height, in cm; length, in cm) will be evaluated during various tests of vertical (Squat Jump and Counter Movement Jump) and horizontal (Single Hop and Triple Hop) jumps.
Jump performances measurement | week 12
  The performance of jumps (height, in cm; length, in cm) will be evaluated during various tests of vertical (Squat Jump and Counter Movement Jump) and horizontal (Single Hop and Triple Hop) jumps.
Postural balance performances measurement | week 6
  The postural balance performance (displacement of the center of pressure, in mm) will be evaluated during a unipodal postural balance test performed on a force platform.
Postural balance performances measurement | week 12
  The postural balance performance (displacement of the center of pressure, in mm) will be evaluated during a unipodal postural balance test performed on a force platform.

CONTACTS AND LOCATIONS:
Overall Officials: Léonard FEASSON, MD PHD, Principal Investigator — Centre Hospitalier de Saint-Etienne; Thomas LAPOLE, PhD, Study Director — Université de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No